CLINICAL TRIAL: NCT00621088
Title: A Prospective Randomised Multicenter Study Comparing the Sliding Hip Screw and the Intertan Nail in Trochanteric and Subtrochanteric Femoral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Kjell Matre, MD, Head of Orthopaedic trauma, Haukeland University Hospital, Department of Orthopaedics, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17972
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Trochanteric and Subtrochanteric Hip Fractures; Treatment With a New Nail or a Sliding Hip Screw

ARMS (1):
- Intertan (Active Comparator)
  Interventions: Procedure: Intertan

INTERVENTIONS:
Procedure: Intertan — Operations performed either with a Sliding Hip Screw or a nail (Intertan)

SUMMARY:
This is a study to compare the new nail "INTERTAN" with a Sliding Hip Screw in treating a specific group of hipfractures (trochanteric and subtrochanteric fractures).

Are there differences in terms of pain, early and late functional mobility and complications between the to implants (and methods of operation)?

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 60 years with a trochanteric or subtrochanteric hip fracture.

Exclusion Criteria:

* Patients with pathologic fractures, patients already included with a fracture on the opposite side.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Early postoperative pain (VAS)(and functional mobility (TUG-test)) | 1 week postoperative

SECONDARY OUTCOMES:
Pain, functional mobility (TUG-test), Harris Hip Score, quality of life (EQ-5D) and complications at discharge from hospital,and at 6 weeks,3 and 12 months postop. | 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Matre, MD, Principal Investigator — Orthopaedic Department, Haukeland University Hospital
Locations (1):
- Orthopaedic dep, Haukeland University Hospital, Bergen, Norway